CLINICAL TRIAL: NCT04271449
Title: tDCS and Prismatic Adaptation: Roles of the Cerebellum and the Primary Motor Cortex in the Transfer of After-effects to a Non-exposed Task.
Brief Title: tDCS and Prismatic Adaptation: Roles of the Cerebellum and the Primary Motor Cortex in the Transfer of After-effects
Acronym: TRANSTIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no inclusion
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 69HCL19_0485; 2019-A02373-54 (Other: ID-RCB)
Record Dates: First submitted 2019-09-10; First posted 2020-02-17 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: prismatic adaptation; tDCS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cerebellum tDCS (Experimental): Cerebellum tDCS arm will be subdivided into two other arms according to the polarity of the stimulation (inhibitory vs excitatory stimulation). These two subgroups will be divided into two other subgroups according the the task exposed during prism exposure (pointing vs throwing).
  Interventions: Device: tDCS (transcranial direct current stimulation)
- Primary motor cortex (Experimental): Primary motor cortex tDCS arm will be subdivided into two other arms according to the polarity of the stimulation (inhibitory vs excitatory stimulation). These two subgroups will be divided into two other subgroups according the the task exposed during prism exposure (pointing vs throwing).
  Interventions: Behavioral: Virtual reality device
- Sham tDCS (Sham Comparator): Sham tDCS arm will serve as a sham comparator for other experimental conditions. This arm will be subdivided into two groups depending on the localisation of the electrodes (cerebellum placement vs primary motor cortex placement).These two subgroups will be divided again in two subgroups depending on the task exposed (pointing vs throwing).
  Interventions: Device: tDCS (transcranial direct current stimulation)

INTERVENTIONS:
Device: tDCS (transcranial direct current stimulation) — Non invasive functional brain stimulation that allows to modulate the excitability of a targeted area (inhibitory or excitatory) thanks to a small current that goes beyond two electrodes. For this arm, the targeted are will be the cerebellum.
  Prismatic googles will also be used in the same way in all groups during prism exposure.
  Arms: Cerebellum tDCS
Behavioral: Virtual reality device — Non invasive functional brain stimulation that allows to modulate the excitability of a targeted area (inhibitory or excitatory) thanks to a small current that goes beyond two electrodes. For this arm, the targeted are will be the cerebellum.
  Prismatic googles will also be used in the same way in all groups during prism exposure.
  Arms: Primary motor cortex
Device: tDCS (transcranial direct current stimulation) — Non invasive functional brain stimulation that allows to modulate the excitability of a targeted area (inhibitory or excitatory) thanks to a small current that goes beyond two electrodes. For this arm, the targeted are will be either the cerebellum or the primary motor cortex, but the stimulation will be turned off after 15 seconds to insure a sham condition.
  Prismatic googles will also be used in the same way in all groups during prism exposure.
  Arms: Sham tDCS

SUMMARY:
Human beings are able to produce precise and smooth movements despite varying demands thank to the nervous system plasticity. Primastic exposure is a method that allows to easily study these sensorimotor plasticity processes in a laboratory context. In a typical protocol, participants wear prismatic goggles that induce a lateral deviation of the visual field while performing a goal directed motor task (e.g. pointing). During the first trials, participants make errors in the direction of the deviation and correct them trial-by-trial. Finally, participants go back to baseline performances after a few dozen of trials. Upon goggles removal, participants make mistakes toward the direction opposition to the initial prismatic deviation. These after-effects reflect adaptive processes that occurred to counteract the perturbation. The way that these after-effects can be transferred to other situations which have not been exposed to the prismatic perturbation bring crucial information about the nature of the processes involved. Additionally, these transfer properties might be of great interest in the field of neuro rehabilitation. In fact, the purpose of therapeutic strategies is to induce compensations that can be transferred to daily life situations.

In previous studies, the investigator showed that expertise on the exposed had a notable influence on transfer properties. However, these studies did not allow to identify the cerebral regions involved in transfer.

The cerebellum is described as a major area implied during motor adaptation and the occurrence of after-effects, while the primary motor cortex might play a crucial role in the formation of motor memory. As such, these two regions are likely to be involved in transfer properties.

The objective of this project is to identify the roles of the cerebellum and the primary motor cortex in the transfer of visuomotor compensations acquired during prism exposure to task that has not been practiced under the perturbation. To do so, the investigator will use transcranial direct current stimulation (tDCS) which is a non-painful and non-invasive functional brain stimulation method. Several groups will be constituted to test if stimulation (inhibitory and excitatory) of the cerebellum or the primary motor on the transfer of prism acquired compensations to a non-exposed task. More precisely, the investigator aim to study the influence of different stimulation modalities (cerebellum vs MA, inhibitory vs excitatory vs sham) on the error reduction during prism exposure, on the amount of after-effects and on the amount on transfer to the non-exposed task.

On a fundamental level, this project will allow a better understanding of the sensorimotor plasticity processes involved to counteract a perturbation and about mechanisms underlying transfer properties. Future results would allows to shed light on the conditions necessary to give rise to transfer as well as the implied brain regions. On longer-term these results will be used to optimize rehabitation strategies in motor function recovery in order to favour the transfer of acquired compensations to daily life situations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Right-handed
* Aged 18 to 70
* Normal or corrected vision
* Signed written informed consent
* Affiliated to a health care organism.

Exclusion Criteria:

* Neurological or psychiatric disorder
* Pregnancy
* Epilepsy antecedents
* Presence of metallic implant, pace maker, cochlear implant, chirurgical brain clip.
* Cognitive disorders
* presence of corrective eyeglasses
* Right upper limb orthopedic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Endpoint lateral errors : lateral distance between the endpoint of the movement and the aimed target assessed by motion capture. | Day 0
  Primary outcome measure will be the endpoint lateral error for each trial, that will be expressed in degrees. The distance between the aimed target and either the final position of the index (pointing trials) or the ball impact (throwing trials) will be recorded with a motion capture system and expressed in centimeters. Then, they will be converted into degrees through trignometric rules, taking in account the distance between the eyes and the target.

SECONDARY OUTCOMES:
Movement velocities of pointing trajectories | Day 0
  Movement velocities (cm/s) at acceleration, velocity and deceleration peaks. Kinematics will be calculated using positions of markers on the arm, recorded by motion capture.
Movement directions of pointing trajectories | Day 0
  Movement movement directions (orientation of velocity vectors in degrees) at acceleration, velocity and deceleration peaks. Kinematics will be calculated using positions of markers on the arm, recorded by motion capture.

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROSSETTI, Principal Investigator — Centre de Recherche en Neuroscience de Lyon INSERM U1028, Equipe ImpAct
Locations (1):
- Centre de Recherche en Neuroscience de Lyon INSERM U1028, Equipe ImpAct, Bron, France